CLINICAL TRIAL: NCT02527746
Title: A Single-Center, Open-Label, Dose-Escalation Phase I Clinical Trial of Recombinant Human Granulocyte Colony Stimulating Factor-Fc Fusion Protein for Injection as an Adjuvant to Chemotherapy in Subjects With Breast Cancer
Brief Title: Study of F-627 in Women With Breast Cancer Receiving Myelotoxic Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EVIVE Biotechnology (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-F-627-CH1
Record Dates: First submitted 2015-07-23; First posted 2015-08-19 (Estimated); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-07

CONDITIONS: Neutropenia; Breast Cancer
MeSH Terms: conditions — Neutropenia; Breast Neoplasms | interventions — EC regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- F-627 80 µg/kg (Experimental): F-627 at the dose of 80 µg/kg administrated by s.c. injection on Day 3 of each cycle for 4 cycles.
  Interventions: Drug: F-627; Drug: EC regimen
- F-627 240 µg/kg (Experimental): F-627 at the dose of 240 µg/kg administrated by s.c. injection on Day 3 of each cycle for 4 cycles.
  Interventions: Drug: F-627; Drug: EC regimen
- F-627 320 µg/kg (Experimental): F-627 at the dose of 320 µg/kg administrated by s.c. injection on Day 3 of each cycle for 4 cycles.
  Interventions: Drug: F-627; Drug: EC regimen

INTERVENTIONS:
Drug: F-627 — F-627 subcutaneous injection on Day 3 of each cycle for 4 cycles. Dose-escalation method was used.
  Other Names: Recombinant Human Granulocyte Colony Stimulating Factor (rh G-CSF) Fc fusion protein
Drug: EC regimen — Epirubicin 100 mg/m^2 (in vein) and Cyclophosphamide 600 mg/m^2 (in vein) on Day 1 of each cycle for 4 cycles.
  Other Names: Epirubicin + Cyclophosphamide

SUMMARY:
A Phase I, dose escalation study to evaluate the safety and pharmacokinetics/pharmacodynamics of F-627 in female breast cancer patients who received up to 4 cycles of Epirubicin and Cyclophosphamide. 18 patients (6 patients each cohort) were assigned to three escalated dose cohorts of 80, 240 and 320 µg/kg.

DETAILED DESCRIPTION:
A Phase I, dose escalation study to evaluate the safety and pharmacokinetics/pharmacodynamics of F-627 in female breast cancer patients receiving 4 cycles of EC (Epirubicin plus Cyclophosphamide) chemotherapy.

18 patients (6 patients each cohort) were assigned to three sequential doses cohort of F-627 at the dose of 80, 240 and 320 µg/kg. The patients received chemotherapy (100 mg/m^2 epirubicin and 600 mg/m^2 cyclophosphamide) administrated by i.v. injection on Day 1 and F-627 by s.c. injection on Day 3 of each cycle for 4 cycles. If no dose-limiting toxicity (DLT) was observed in 6 patients during first cycle, the next cohort was escalated.

Blood samples were collected for completed blood counts with differential, serum F-627 concentration and safety evaluation at different point following F-672 injection.

The decision to proceed to the next higher dose was made jointly by the sponsor's medical expert and the investigator based upon the review of safety data in the first cycle treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old.
2. Female postoperative breast cancer patients who require adjuvant chemotherapy, and are planned to receive 4 cycles of EC chemotherapy;
3. East Cooperative Oncology Group (ECOG) performance 0-1.
4. Absolute neutrophil count (ANC) ≥ 2.0 × 10^9/L, hemoglobin (Hb) ≥ 11.0 g/dl, and platelets (PLT) ≥ 100 × 10^9/L prior to chemotherapy.
5. Hepatic and renal function within the normal range;.
6. Left ventricular ejection fraction (LVEF) > 50%.
7. Willing to sign the informed consent form and able to comply with protocol requirements

Exclusion Criteria:

1. Women in pregnancy or breastfeeding; Women of child-bearing potential have a positive pregnancy test result prior to the first dose;
2. Life expectancy less than 12 months;
3. Radiation therapy within 4 weeks prior to enrollment;
4. Breast cancer patients who have received neoadjuvant chemotherapy before radical mastectomy;
5. Prior bone marrow or stem cell transplant;
6. With other malignant tumors other than breast cancer;
7. Have received granulocyte colony stimulating factor (G-CSF) treatment within 6 weeks prior to enrollment;
8. Diagnosed with acute congestive heart failure, cardiomyopathy, or myocardial infarction by clinical diagnosis, electrocardiograph (ECG) or other approaches;
9. With any disease that may cause splenomegaly;
10. With acute infection, chronic active Hepatitis B within 1 year (unless patients tested negative for HBsAg prior to enrollment), or Hepatitis C;
11. History of tuberculosis (TB); history of TB exposure, unless negative for tuberculin test; TB patients undergoing treatment; or suspected TB evaluated by chest x-ray;
12. Known human immunodeficiency virus (HIV) positive or acquired immune deficiency syndrome (AIDS);
13. With sickle cell anemia;
14. With alcohol or drug abuse that may affect the compliance with the study;
15. With known hypersensitivity to E. coli derived proteins, G-CSF, or excipients;
16. Has received any other investigational drug within 4 weeks prior to enrollment;
17. Patients with diseases or symptoms unsuitable for participating in the clinical trial based on the investigator's judgment;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junning Cao, Professor, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- F-627 80 µg/kg: F-627 at the dose of 80 µg/kg administrated by s.c. injection on Day 3 of each cycle for 4 cycles.
  F-627: F-627 subcutaneous injection on Day 3 of each cycle for 4 cycles. Dose-escalation method was used.
  Epirubicin+Cyclophosphamide (EC) regimen: Epirubicin 100 mg/m^2 (in vein) and Cyclophosphamide 600 mg/m^2 (in vein) on Day 1 of each cycle for 4 cycles.
Period: Overall Study
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (9.50) | 49.0 (4.90) | 54.5 (11.20) | 49.8 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 18
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Safety of F-627 for Injection in the Treatment of Female Postoperative Patients With Breast Cancer Who Require Adjuvant Chemotherapy.
Description: Safety endpoints include incidence rate and severity of adverse events (AEs), laboratory measurements, physical examinations, vital signs, and performance status. Severity of AEs were assessed according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 4.03 criteria.
Time Frame: Up to 4 cycles (about 84 days)
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
Participants
  Number of subjects who reported AEs | 6 | 6 | 6
  Number of subjects who reported TEAEs | 6 | 6 | 6
  Number of subjects who reported investigational drug-related TEAEs | 3 | 3 | 4
  Number of subjects who reported grade 3 or greater TEAEs | 6 | 4 | 5
  Number of subjects who reported grade 3 or greater investigational drug-related TEAEs | 0 | 0 | 0
  Number of subjects who reported TEAEs leading to permanent discontinuation | 0 | 0 | 0
  Number of subjects who reported serious adverse events (SAEs) | 0 | 1 | 0
  Number of subjects who reported of investigational drug-related serious adverse events (SAEs) | 0 | 0 | 0

2. Primary Outcome: Tolerability (Dose-limiting Toxicity) of F-627 for Injection in the Treatment of Female Postoperative Patients With Breast Cancer Who Require Adjuvant Chemotherapy.
Description: Tolerability should be assessed by dose-limiting toxicity (DLT). DLT is defined as any grade 3 or greater adverse event related to the investigational drug that observed in cycle 1 (21 days).
Time Frame: Up to 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
Participants | 0 | 0 | 0

3. Secondary Outcome: T1/2 of F-627 in Each Dose Cohort in Cycle 1 and Cycle 3
Description: There are a total of 13 blood sampling time points in each cycle: pre-dose and 2, 6, 12, 24, 36, 48, 72, 96, 120, 144, 192, and 240 hr after dosing. Two additional sampling time points, 312 and 432 hr after dosing, are included for the 320 μg/kg cohort. Serum drug concentrations of F-627 at different time points will be determined using enzyme linked immunosorbent assay (ELISA).
Time Frame: Cycle 1 and cycle 3 (each cycle was about 21 days)
Measure: Median (Full Range); unit: hours
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
hours
  Cycle 1 T1/2 | 49.88 [38.71 to 76.67] | 34.71 [19.39 to 86.05] | 56.37 [31.14 to 112.95]
  Cycle 3 T1/2 | 73.44 [55.28 to 210.58] | 61.95 [45.79 to 131.79] | 44.58 [31.05 to 109.27]

4. Secondary Outcome: Cmax of F-627 in Each Dose Cohort in Cycle 1 and Cycle 3
Description: There are a total of 13 blood sampling time points in each cycle: pre-dose and 2, 6, 12, 24, 36, 48, 72, 96, 120, 144, 192, and 240 hr after dosing. Two additional sampling time points, 312 and 432 hr after dosing, are included for the 320 μg/kg cohort. Serum drug concentrations of F-627 at different time points will be determined using ELISA.
Time Frame: Cycle 1 and cycle 3 (each cycle was about 21 days)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Cycle 1 Cmax | 25.77 (7.22) | 226.80 (101.70) | 192.87 (76.06)
  Cycle 3 Cmax | 29.06 (27.53) | 73.09 (26.16) | 85.17 (46.71)

5. Secondary Outcome: Tmax of F-627 in Each Dose Cohort in Cycle 1 and Cycle 3
Description: as for outcome 4
Time Frame: Cycle 1 and cycle 3 (each cycle was about 21 days)
Measure: Median (Full Range); unit: hours
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
hours
  Cycle 1 Tmax | 24 [12.00 to 36.00] | 36.00 [12.00 to 48.00] | 48.15 [24.30 to 120.20]
  Cycle 3 Tmax | 12.00 [5.80 to 12.00] | 9.10 [6.00 to 24.20] | 12.00 [11.50 to 12.00]

6. Secondary Outcome: Area Under Curve (AUC)0-t of F-627 in Each Dose Cohort in Cycle 1 and Cycle 3
Description: as for outcome 4
Time Frame: Cycle 1 and cycle 3 (each cycle was about 21 days)
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL
  Cycle 1 Area Under Curve (AUC) | 2477.75 (661.64) | 15230.79 (4851.43) | 19858.38 (7503.75)
  Cycle 3 Area Under Curve (AUC) | 1586.35 (632.57) | 4347.35 (2135.28) | 6556.98 (2683.3)

7. Secondary Outcome: Vz/F of F-627 in Each Dose Cohort in Cycle 1 and Cycle 3
Description: as for outcome 4
Time Frame: Cycle 1 and cycle 3 (each cycle was about 21 days)
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
mL/kg
  Cycle 1 Vz/F | 2457.22 (975.35) | 1238.80 (1336.92) | 1597.02 (646.10)
  Cycle 3 Vz/F | 6196.75 (3477.13) | 6132.23 (2997.45) | 4079.81 (2189.98)

8. Secondary Outcome: Cl/F of F-627 in Each Dose Cohort in Cycle 1 and Cycle 3
Description: as for outcome 4
Time Frame: Cycle 1 and cycle 3 (each cycle was about 21 days)
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
mL/h/kg
  Cycle 1 Cl/F | 31.34 (7.14) | 17.11 (6.94) | 18.89 (9.78)
  Cycle 3 Cl/F | 45.41 (16.47) | 62.45 (35.67) | 56.38 (26.24)

9. Secondary Outcome: Mean Residence Time (MRT)0-t of F-627 in Each Dose Cohort in Cycle 1 and Cycle 3
Description: as for outcome 4
Time Frame: Cycle 1 and cycle 3 (each cycle was about 21 days)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
hours
  Cycle 1 Mean residence time (MRT) | 86.85 (11.70) | 61.98 (18.90) | 88.69 (18.73)
  Cycle 3 Mean residence time (MRT) | 87.08 (18.97) | 75.61 (7.44) | 96.29 (25.61)

10. Secondary Outcome: Percentage of Subjects With Grade 3 or 4 Neutropenia (< 1.0 × 10^9/L)
Description: For cycle 1, starting on day 3, oral temperature measurement and routine blood test (including ANC) will be performed daily until ANC recovers to no less than 1.0 × 10^9/L from nadir, and once every 3 days thereafter until the next cycle; for chemotherapy cycles 2-4 (day 3-day 21 of each chemotherapy cycle, i.e., day 24-day 84 of the study), starting on day 3, oral temperature measurement and routine blood test will be performed every other day until ANC recovers to no less than 1.0 × 10^9/L from nadir, and once every 3 days thereafter until the next cycle.
Time Frame: Up to 4 cycles (84 days)
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
Participants
  Percentage of subjects with grade 3 or 4 neutropenia (%) in cycle 1 | 6 | 3 | 5
  Percentage of subjects with grade 3 or 4 neutropenia (%) in cycle 2 | 0 | 2 | 0
  Percentage of subjects with grade 3 or 4 neutropenia (%) in cycle 3 | 3 | 2 | 1
  Percentage of subjects with grade 3 or 4 neutropenia (%) in cycle 4 | 4 | 2 | 2

11. Secondary Outcome: Percentage of Subjects With Grade 4 Neutropenia (< 0.5 × 10^9/L)
Description: as for outcome 10
Time Frame: Up to 4 cycles (84 days)
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
Participants
  Percentage of subjects with grade 4 neutropenia (%) in cycle 1 | 3 | 3 | 2
  Percentage of subjects with grade 4 neutropenia (%) in cycle 2 | 0 | 0 | 0
  Percentage of subjects with grade 4 neutropenia (%) in cycle 3 | 0 | 1 | 0
  Percentage of subjects with grade 4 neutropenia (%) in cycle 4 | 2 | 2 | 0

12. Secondary Outcome: Duration of Absolute Neutrophil Count (ANC)< 0.5 × 10^9/L (Days)
Description: as for outcome 10
Time Frame: Up to 4 cycles (84 days)
Population: This outcome measure applies to all participants with a valid ANC level, regardless of whether the ANC level is less than 0.5 × 10^9/L.
  The value of 0 represents the participant experienced 0 days with ANC < 0.5 × 10^9/L (days).
  The Number of Participants Analyzed for *each* Row is the same with the Overall Number of Participants Analyzed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
days
  Duration of ANC < 0.5 × 10^9/L (days) in cycle 1 | 0.8 (0.98) | 1.2 (1.33) | 0.5 (0.84)
  Duration of ANC < 0.5 × 10^9/L (days) in cycle 2 | 0 (0) | 0 (0) | 0 (0)
  Duration of ANC < 0.5 × 10^9/L (days) in cycle 3 | 0 (0) | 0.2 (0.41) | 0 (0)
  Duration of ANC < 0.5 × 10^9/L (days) in cycle 4 | 0.3 (0.52) | 0.3 (0.52) | 0 (0)

13. Secondary Outcome: Duration of Absolute Neutrophil Count (ANC)< 1.0 × 10^9/L (Days)
Description: as for outcome 10
Time Frame: Up to 4 cycles (84 days)
Population: This outcome measure applies to all participants with a valid ANC level, regardless of whether the ANC level is less than 1.0 × 10^9/L.
  The value of 0 represents the participant experienced 0 days with ANC < 1.0 × 10^9/L (days).
  The Number of Participants Analyzed for *each* Row is the same with the Overall Number of Participants Analyzed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
days
  Duration of ANC < 1.0 × 10^9/L (days) in cycle 1 | 2.8 (0.75) | 1.5 (1.76) | 1.5 (1.05)
  Duration of ANC < 1.0 × 10^9/L (days) in cycle 2 | 0 (0) | 0.3 (0.52) | 0 (0)
  Duration of ANC < 1.0 × 10^9/L (days) in cycle 3 | 0.7 (0.82) | 0.3 (0.52) | 0.2 (0.41)
  Duration of ANC < 1.0 × 10^9/L (days) in cycle 4 | 1.0 (1.10) | 0.7 (1.03) | 0.5 (0.84)

14. Secondary Outcome: Absolute Neutrophil Count (ANC) Nadir (10^9 Cells/L)
Description: as for outcome 10
Time Frame: Up to 4 cycles (84 days)
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
10^9 cells/L
  ANC Nadir (10^9/L) in cycle 1 | 0.50 (0.352) | 0.90 (1.056) | 0.72 (0.360)
  ANC Nadir (10^9/L) in cycle 2 | 1.57 (0.339) | 1.97 (1.193) | 2.33 (0.841)
  ANC Nadir (10^9/L) in cycle 3 | 1.52 (0.833) | 2.42 (2.260) | 2.20 (0.976)
  ANC Nadir (10^9/L) in cycle 4 | 0.87 (0.589) | 2.02 (1.551) | 1.63 (0.862)

15. Secondary Outcome: Time (Days) of Absolute Neutrophil Count (ANC) Recovered to 1.0 × 10^9/L From Nadir
Description: as for outcome 10
Time Frame: Up to 4 cycles (84 days)
Population: This outcome measure applies to all participants with a valid ANC level, regardless of whether the ANC level is less than 1.0 × 10^9/L.
  The value of 0 represents the participant experienced 0 days with ANC recovered to 1.0 × 10^9/L from nadir.
  The Number of Participants Analyzed for *each* Row is the same with the Overall Number of Participants Analyzed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
Number analyzed (Participants) | 6 | 6 | 6
days
  Time (days) of ANC recovered to 1.0 × 10^9/L from nadir in cycle 1 | 2.5 (0.55) | 1.2 (1.47) | 1.0 (0.63)
  Time (days) of ANC recovered to 1.0 × 10^9/L from nadir in cycle 2 | 0.0 (0.00) | 0.7 (1.03) | 0.0 (0.00)
  Time (days) of ANC recovered to 1.0 × 10^9/L from nadir in cycle 3 | 1.3 (1.63) | 0.7 (1.03) | 0.3 (0.82)
  Time (days) of ANC recovered to 1.0 × 10^9/L from nadir in cycle 4 | 1.0 (0.89) | 0.7 (1.03) | 0.7 (1.03)

ADVERSE EVENTS:
Time Frame: From the first treatment of chemotherapy until the end of study at Day 84
Description: Summary of Adverse Events includes only those participants who received at least one dose of investigational product
Arm/Group | F-627 80 µg/kg | F-627 240 µg/kg | F-627 320 µg/kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F-627 80 µg/kg (N=6) | F-627 240 µg/kg (N=6) | F-627 320 µg/kg (N=6)
febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F-627 80 µg/kg (N=6) | F-627 240 µg/kg (N=6) | F-627 320 µg/kg (N=6)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 2 (3) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (5)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 6 (14) | 6 (16) | 6 (19)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 6 (71) | 6 (41) | 6 (32)
Alanine Aminotransferase Increased (Investigations) | 1 (3) | 1 (2) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
White blood cells urine positive (Investigations) | 2 (2) | 0 (0) | 3 (3)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 3 (4) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 6 (56) | 5 (33) | 6 (23)
Aspartate Aminotransferase Increased (Investigations) | 1 (3) | 1 (2) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 1 (1) | 2 (2)
Haemoglobin Decreased (Investigations) | 6 (32) | 6 (64) | 4 (31)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 2 (9) | 4 (19) | 5 (21)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Wound Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (10) | 5 (9) | 6 (8)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 5 (9) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (9) | 5 (13) | 6 (13)
Effusion (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (12) | 0 (0) | 0 (0)
Gingival Bleeding (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Gingival Swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (17) | 5 (15) | 5 (16)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 3 (5) | 0 (0) | 2 (3)
Mouth Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (19) | 5 (20) | 5 (14)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival inflammation (Gastrointestinal disorders) | 2 (4) | 1 (1) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 5 (6) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2013-05-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT02527746/Prot_000.pdf
  • Statistical Analysis Plan (2013-12-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT02527746/SAP_001.pdf